CLINICAL TRIAL: NCT04174456
Title: Olmesartan Effect on Myocardial Viability of Patients With Dilated Cardiomyopathy
Brief Title: Combination of Olmesartan Effect on Myocardial Viability of Patients With Dilated Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Kyungil Park, Associate professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-215
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olmesartan group (Experimental): olmesartan 20mg once daily with rosuvastatin 5mg once a day for 6-month
  Interventions: Diagnostic Test: FDG PET
- Valsartan group (Active Comparator): valsartan 40mg twice daily with rosuvastatin 5mg once a day for 6-month
  Interventions: Diagnostic Test: FDG PET

INTERVENTIONS:
Diagnostic Test: FDG PET — baseline and 6-month follow-up FDG PET

SUMMARY:
The study proceeds with prospective, randomized, open and controlled clinical trials. The subject of the investigator's study was the first patient diagnosed with dilated cardiomyopathy. Subjects who agreed to participate in the study and were determined to meet the selection / exclusion criteria were randomly assigned to each group, and the experimental group was treated with 20 mg of olmesartan and 5 mg of rosuvastatin for 6 months, and the control group is treated with 40 mg of valsartan and 5 mg of rosuvastatin.

DETAILED DESCRIPTION:
Myocardial viability plays an important role in improving the function of the heart. To date, the most reproducible and objective method has been established as a method or tool for assessing myocardial viability.

Olmesartan is known to have the strongest inhibitory ability of angiotensin receptors compared with other angiotensin receptor binding inhibitors. Research has been reported that statin drugs may help improve vascular endothelial function, and several researchers have suggested that these mechanisms may affect the improvement of myocardial survival. In addition, studies have shown that angiotensin receptor binding inhibitors and statins may improve left ventricular function in patients with left ventricular function. However, since the studies did not assess myocardial survival, the mechanisms could not be clearly identified.

The purpose of this study is to investigate the effect of olmesartan on myocardial survival in patients with dilated cardiomyopathy who have left ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* dilated cardiomyopathy

Exclusion Criteria:

* contraindication to angiotensin receptor blocker
* cardiogenic shock
* sensitive to rosuvastatin
* liver cirrhosis more than Child class B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of glucose metabolism | 6 month
  data from fludeoxyglucose positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Kyungil PARK, Study Director — Dong-A University Hospital
Locations (1):
- Department of Internal Medicine,Dong-A University College of Medicine, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
We don't have any plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Jo S, Park K, Choi JH, Sohn CB, Kim J, Kwon YS, Kim SH, Park TH. A Comparison Study of Olmesartan and Valsartan Effects on Myocardial Metabolism in Patients With Dilated Cardiomyopathy: the OVOID Trial. J Am Heart Assoc. 2025 Jul;14(13):e041406. doi: 10.1161/JAHA.125.041406. Epub 2025 Jun 27. PMID 40576039
- [Derived] Jo S, Moon H, Park K, Sohn CB, Kim J, Kwon YS, Kim SH. Design and rationale for a comparison study of Olmesartan and Valsartan On myocardial metabolism In patients with Dilated cardiomyopathy (OVOID) trial: study protocol for a randomized controlled trial. Trials. 2022 Jan 15;23(1):36. doi: 10.1186/s13063-021-05970-7. PMID 35033178